CLINICAL TRIAL: NCT00209196
Title: Health Behaviors and Quality of Life in Pediatric Solid Organ Transplant Recipients
Brief Title: Quality of Life in Pediatric Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Laura L. Mee, Psychologist, Emory University
Other Study IDs: IRB00045836
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Kidney Transplantation; Liver Transplantation; Heart Transplantation; Lung Transplantation; Heart-Lung Transplantation
Keywords: pediatric; transplantation; psychosocial; kidney transplant recipient; liver transplant recipient; heart transplant recipient; lung transplant recipient; heart-lung transplant recipient

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pediatric solid organ transplants: Adherence to medical regimens refers to what degree a patient chooses to follow the advice given by his/her healthcare provider.More recently, researchers have started to look at adherence with children who have undergone solid organ transplantation. This is because about 50% of these children are to some degree non-adherent with their medical regimen. This comes at a costly price as ongoing non-adherence in pediatric transplant can lead to the child's body rejecting the new organ and even death. This study has been designed to look at the reasons that pediatric patients may choose to be non-adherent.

SUMMARY:
Adherence to medical regimens refers to what degree a patient chooses to follow the advice given by his/her healthcare provider. Good adherence typically involves behaviors such as the patient taking medication as directed and going to scheduled clinic appointments. As many patients often do not follow the advice of doctors as closely as suggested, many researchers have tried to find out the reasons behind patients being "non-adherent." This research has looked at medical conditions such as diabetes, cystic fibrosis, and asthma. More recently, researchers have started to look at adherence with children who have undergone solid organ transplantation. This is because about 50% of these children are to some degree non-adherent with their medical regimen. This comes at a costly price as ongoing non-adherence in pediatric transplant can lead to the child's body rejecting the new organ and even death. This study has been designed to look at the reasons that pediatric patients may choose to be non-adherent. This study will look at issues related to the patient (e.g., age, family support), related to the disease and regimen (e.g., length of illness, how complicated the regimen is), related to the medication (e.g., taste, side effects), related to their mind (e.g., memory problems, confusion), and related to their emotions (e.g., being depressed, anxious). The investigators will be looking at each regimen-related behavior, such as attending clinic appointments and will be asking each family about any barriers that make it difficult. The investigators hope that knowing these barriers will help them make interventions that fit the specific issues that each patient faces. Ultimately, doctors, transplant coordinators, and psychological professionals will be able to use this information to intervene early with families who report barriers that impact adherence.

DETAILED DESCRIPTION:
This study will involve approximately 100 parents of pediatric patients who have received a solid organ transplant at Children's Healthcare of Atlanta (CHOA) between January 1st, 1988 and December 31st, 2004. Within this sample, pediatric patients who are 11-18 years of age will be invited to participate in a separate component of the project, involving approximately 50 adolescents.

ELIGIBILITY CRITERIA:

For a parent to participate in this study the child must have had a solid organ transplant at CHOA, patient is 5-18 years of age, patient lives with the parent(s) in the home, and informed consent can be obtained. For a child to participate in this study, the child must have had a solid organ transplant at CHOA, patient is 11-18 years of age, patient lives with the parent(s) in the home, and informed assent can be obtained. Family exclusionary criteria are as follows:

* patient has not lived with parent for at least 6 months
* patient's medical records are not accessible through the CHOA system.

All participants will be referred by the respective transplant coordinator or one of the physicians in this study. Parents will be provided with the findings upon request and referrals for psychological services will be made as necessary.

RECRUITMENT:

To recruit participants for the proposed study, children and adolescents who received a solid organ transplant at CHOA between January 1st, 1988 and December 31st, 2004 will be identified by the transplant coordinators or physician for each solid organ. Although multiple methods of recruitment will be used, each family will only be contacted once.

Clinic recruitment with the investigator present:

Any patient family who is scheduled for an upcoming clinic visit will be approached by the transplant coordinator or other clinic-affiliated individual. The investigation will be briefly described and interest in participating will be solicited.

The parent will sign a letter of interest stating either:

1. They are interested in learning more. The form will also ask them to provide contact information (home address and telephone number) or
2. They are not interested and do not want to be contacted further.

Only letters indicating interest will be given to investigators. If a family signs the letter indicating interest, an investigator present at clinic will approach the family to describe the investigation and obtain consent/assent. The family will have the option to:

1. conduct the interview during the present clinic visit,
2. schedule a future time to conduct the interview at the clinic, or
3. conduct the interview via telephone.

Clinic recruitment with the investigator not present:

If an investigator is not present at the clinic, the transplant coordinator or other clinic-affiliated individual will give the letters indicating interest to an investigator to contact the family via telephone to describe the study. If after the telephone conversation, a parent is interested in participating, 2 copies of the consent form will be sent to the parent's home with a self-addressed envelope to return one signed copy. Following receipt of this form, the parent will be contacted to schedule either:

1. an interview at the clinic or
2. an interview via telephone.

Mail recruitment:

Any patient family who is not scheduled for an upcoming clinic visit will be contacted via mail from the transplant coordinator and transplant physician. The letter will briefly describe the investigation and a letter of interest will be included. Included will be a postage-paid envelope to return directly to the transplant team. The transplant coordinator or other clinic-affiliated individual will give the letters indicating interest to an investigator to contact the family via telephone to describe the study. If after the telephone conversation, a parent would like to participate, 2 copies of the consent form will be sent to the parent's home with a self-addressed envelope to return one signed copy to the investigator. Following receipt of this form, the parent will be contacted to schedule either:

1. an interview at the clinic or
2. an interview via telephone.

Telephone recruitment:

If a parent is not seen in the clinic and does not return a letter of interest, the transplant coordinator or other clinic affiliated individual will call the family to briefly describe the investigation and obtain verbal consent for an investigator to contact them via telephone. If they indicate that they are not interested in participating, they will not be contacted further. If a parent verbally consents to being contacted to learn more about the study, an investigator will contact the family via telephone. If after the telephone conversation, a parent would like to participate, 2 copies of the consent form will be sent to the parent's home with a self-addressed envelope to return one signed copy to the investigator. Following receipt of this form, the parent will be contacted to schedule either:

1. an interview at the clinic or
2. an interview via telephone.

If the family is called three times with no success in reaching them, this will be considered passive refusal and will not be contacted further.

INTERVIEW PROCEDURE:

The interview with each parent will consist of verbal consent and verbal administration of the PEDS-TX Survey, Parent Version 1.0, the Medical Adherence Measure (MAM), the Child Health Questionnaire-Parent Form 50 (CHQ-PF50), the SF-12 Health Survey (SF-12), the Family Relationship Index (FRI), and demographic questions. The interview with each participating adolescent patient will consist of verbal assent and the PEDS-TX Survey, Adolescent Version 1.0, the Medical Adherence Measure (MAM), the Child Health Questionnaire-Child Form 80 (CHQ-CF80), the Adolescent Risk Taking Survey (ARTS), and the Family Relationship Index (FRI). Each interview will be conducted by research assistants and/or graduate students in psychology. They will be trained in all research procedures by the principal investigator. Training will include observed practice of procedures and skills taught, focused on building rapport with and being sensitive to parents and patients with solid organ transplants, verbally administering the assessment questionnaires in an accurate and comfortable manner, giving answers to questions from parents and patients in an instructive manner that do not bias the research, and lastly, being culturally and socioeconomically sensitive when greeting and interviewing families.

The data for this study will likely be obtained over a 6-9 month period, with data from a specific parent and adolescent patient pair occurring within less than a week period (ideally during the same phone call). Each interview will last approximately 45-75 minutes.

MEASURES:

The measures for this investigation are as follows:

* Clinician Derived Measures

  * Medical Record Review
  * Prescription Refill records
* Self-Report Measures
* Demographic Information
* PEDS-TX Survey, Parent and Adolescent Version 1.0
* Medical Adherence Measure
* Child Health Questionnaire-Parent Form 50
* SF-12 Health Survey
* Family Relationship Index
* Child Health Questionnaire-Child Form 80
* Adolescent Risk Taking Survey.

ELIGIBILITY:
Inclusion Criteria:

* Solid organ transplant at Children's Healthcare of Atlanta (CHOA)
* 11-18 years of age
* Lives with the parents in the home
* Signed informed consent

Exclusion Criteria:

* Has not lived with parent for at least 6 months
* Medical records are not accessible through the CHOA system

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male or female Patients at Children's Healthcare of Atlanta Patients at least 11 years old and living at home for 6 months Solid organ transplant patients between 1.1.1988 and 12.31.2004
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2005-05; Primary Completion 2007-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pediatric Quality of Life Measure (Peds QL) | up to one year
  paper questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mee, PhD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States